CLINICAL TRIAL: NCT03373019
Title: A Non-randomized, Open-label, Phase II Study of Chidamide Combined With R-GDP in Treating Patients With Relapsed or Refractory Diffuse Large B-cell Lymphoma (DLBCL) Not Suitable for Transplantation
Brief Title: Chidamide Combined With R-GDP in Treating Patients With Relapsed or Refractory Diffuse Large B-cell Lymphoma (DLBCL)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Kai Xue, MD, Dr, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-RD1
Record Dates: First submitted 2017-11-30; First posted 2017-12-14 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Chidamide; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Neoplasm by Histology; Neoplasms; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases; Lymphoma, Non-Hodgkin; Cyclophosphamide; Rituximab; Gemcitabine; Cisplatin; Dexamethasone; HDAC Inhibitor
Keywords: chidamide; R-GDP; diffuse large B-cell lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Neoplasms; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chidamide combined with R-GDP (Experimental): Chidamide: 30mg,PO,biw one week before cycle 1 treatment rituximab 375 mg/m2,ivgtt D0 gemcitabine 1000mg/m2 iv D1,8 dexamethasone 40mg, iv D1-4, cisplatin 25mg/m2 iv D1-4 chidamide :20mg PO Biw, 2 week on , 1 week off
  Interventions: Drug: Chidamide combined with R-GDP

INTERVENTIONS:
Drug: Chidamide combined with R-GDP — Chidamide: 30mg,PO,biw one week before cycle 1 treatment rituximab 375 mg/m2,ivgtt D0 gemcitabine 1000mg/m2 iv D1,8 dexamethasone 40mg, iv D1-4, cisplatin 25mg/m2 iv D1-4 chidamide :20mg PO Biw, 2 week on , 1 week off

SUMMARY:
The goal of this clinical trial is to evaluate therapeutic efficacy of Chidamide combined with R-GDP （rituximab/gemcitabine/dexamethasone/cisplatin）in treating Patients with relapsed or refractory Diffuse Large B-cell Lymphoma (DLBCL) not suitable for transplantation.

DETAILED DESCRIPTION:
The treatment outcome of patients with relapsed or refractory Diffuse Large B-cell Lymphoma (DLBCL) are not satisfactory especially for those not suitable for transplantation. One of main reason is chemotherapy resistance. The investigators conducted this study to evaluate the efficacy of Chidamide combined with R-GDP(rituximab/gemcitabine/dexamethasone/cisplatin) in treating patients with relapsed or refractory Diffuse Large B-cell Lymphoma (DLBCL) not suitable for transplantation. Chidamide is a novel benzamide type of subtype-selective histone deacetylase (HDAC) inhibitor. It has been approved by China Food and Drug Administration (CFDA) for treatment of relapsed or refractory peripheral T-cell lymphoma (PTCL) in Chinese population. The investigators' pre-clinical data suggested that this agent might be also efficient in the treatment of relapsed/refractory B cell lymphoma. In this open-label, non-randomized, phase II study, the investigators aimed to observe the efficacy and safety of chidamide combined with R-GDP in patients with relapsed or refractory Diffuse Large B-cell Lymphoma (DLBCL) not suitable for transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Ages: 18-75 years old
2. Relapsed or refractory Diffuse Large B-cell Lymphoma (DLBCL) previous treated with standard chemoimmunotherapy
3. Not willing or not suitable for hematopoietic stem cell transplantation (HSCT)
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) index < 2
5. Informed consent available
6. Life expectancy of more than 3 months;
7. Ultrasonic cardiogram showed left ventricle ejection fraction ≥ 50%, EKG showed on signs of myocardial ischemia, with no previous arrhythmia which need pharmacological intervention.
8. Bone marrow function: ANC ≥ 1.5 × 109/L, PLT ≥ 100 × 109/L, Hb ≥ 80g/L;
9. Liver function: total bilirubin, ALT and AST were <1.5 × UNL (the upper limit of normal value)
10. Renal function: Cr<1.5 × UNL and creatinine clearance > 50ml/min

Exclusion Criteria:

1. Prior history of treatment of HDAC inhibitor.
2. Plan of HSCT in the future
3. Significant pericardial effusion showed by chest CT scan
4. Prior history of other cancers except treated cervical or basal cell skin carcinoma, organ transplantation
5. Syphilis or human immunodeficiency virus (HIV) infection
6. Pregnant or lactating women
7. History of organ transplantation
8. Serious active infections (including hepatitis)
9. Serious neurological or psychiatric history, including dementia or epilepsy.

Termination criteria:

1. Withdrew consent
2. Researchers think it is necessary to terminate the study;
3. Disease progression or death;
4. Poor compliance
5. Subclinical or clinical cardiac toxicity;
6. Unable to continue treatment because of severe toxicity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2017-12-21 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 6 weeks
  overall response rate

SECONDARY OUTCOMES:
CR | 6 weeks
  complete response
OS | 3 years
  overall survival
3 year PFS | 3 years
  3 year progression free survival
adverse event | throughout the treatment period，up to 6 months
  adverse event related to treatment

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Kai Xue, Shanghai, Shanghai Municipality
  - Kai Xue, Shanghai

IPD SHARING:
Plan to Share IPD: No